CLINICAL TRIAL: NCT00026858
Title: Total Body Irradiation for Bone Marrow Transplants: Collaborative Efforts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950003; 95-C-0003
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-11

CONDITIONS: Neoplasm
Keywords: Bone Marrow Transplantation; Leukemia; Breast Cancer; Multiple Myeloma; Total Body Irradiation
MeSH Terms: conditions — Neoplasms; Leukemia; Breast Neoplasms; Multiple Myeloma | interventions — Intersectoral Collaboration

INTERVENTIONS:
Behavioral: collaboration

SUMMARY:
Most bone marrow transplantations for malignant and non-malignant disease include whole body irradiation. Techniques for administering that treatment, including patient positioning, lung and soft tissue compensation, dose rate, total dose and fractionation differ between institutions. These differences are optimized at each institution to limit toxicity and maximize therapeutic outcome.

Technically complex procedures such as total body radiation are subject to equipment failures. Such failures mid-treatment could be catastrophic to the patient, since therapy must be timely and compatible therapy may not be available elsewhere in the community. The purpose of this protocol is to provide backup between George Washington University Medical Center and the Radiation Oncology Branch of the NCI to allow for orderly, safe, and compatible therapies in the event of equipment failure; or replacement of a linear accelerator or any other malfunctioning equipment necessary to deliver TBI; or any emergent situation.

DETAILED DESCRIPTION:
Most bone marrow transplantations for malignant and non-malignant disease include whole body irradiation. Techniques for administering that treatment, including patient positioning, lung and soft tissue compensation, dose rate, total dose and fractionation differ between institutions. These differences are optimized at each institution to limit toxicity and maximize therapeutic outcome.

Technically complex procedures such as total body radiation are subject to equipment failures. Such failures mid-treatment could be catastrophic to the patient, since therapy must be timely and compatible therapy may not be available elsewhere in the community. The purpose of this protocol is to provide backup between George Washington University Medical Center and the Radiation Oncology Branch of the NCI to allow for orderly, safe, and compatible therapies in the event of equipment failure; or replacement of a linear accelerator or any other malfunctioning equipment necessary to deliver TBI; or any emergent situation.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must sign informed consent.

Supporting institution physicians must agree that therapy is appropriate and safe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1994-10; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Tarbell NJ, Amato DA, Down JD, Mauch P, Hellman S. Fractionation and dose rate effects in mice: a model for bone marrow transplantation in man. Int J Radiat Oncol Biol Phys. 1987 Jul;13(7):1065-9. doi: 10.1016/0360-3016(87)90046-0. PMID 3298176
- [Background] Thomas E, Storb R, Clift RA, Fefer A, Johnson FL, Neiman PE, Lerner KG, Glucksberg H, Buckner CD. Bone-marrow transplantation (first of two parts). N Engl J Med. 1975 Apr 17;292(16):832-43. doi: 10.1056/NEJM197504172921605. No abstract available. PMID 234595
- [Background] Champlin RE, Goldman JM, Gale RP. Bone marrow transplantation in chronic myelogenous leukemia. Semin Hematol. 1988 Jan;25(1):74-80. No abstract available. PMID 3279516